CLINICAL TRIAL: NCT03612908
Title: TSHβX1 Splice Variant Expression and D2 Thr92Ala Polymorphism Analysis in Pregnant Women With Thyroid Diseases
Brief Title: TSHβX1 and D2 THR92ALA in Pregnancy
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other); Ciprés Grupo Médico CGM SC (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: 217B500402016054
Record Dates: First submitted 2018-07-20; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Pregnancy Related; Hypothyroidism; Hyperthyroidism
Keywords: Hyperthyroidism; Polymorphism; TSHβX1; D2 THR92ALA; Hypothyroidism
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normothyroid pregnant women: Healthy pregnant women with the TSH serum values within the recommended ranged per trimester of pregnancy.
- Patients with a thyroid disease: Patients with a thyroid disease named hypothyroidism or hyperthyroidism.

SUMMARY:
Thyroid diseases are pathologies that frequently affect pregnant women causing serious complications. This current research aims to find out whether the expression of TSHβX1 splice variant and D2 Thr92Ala polymorphism in the DIO2 gene are associated with thyroid disease in Mexican pregnant women.

DETAILED DESCRIPTION:
Deiodinase 2 (DIO2) is a selenoenzyme responsible for the deiodination of T4 to T3, which makes it crucial for the proper functioning of thyroid hormones. Polymorphisms of DIO2 alters the enzymatic function. In addition, the Ala92Ala genotype was reported to be related with a reduction in the placental activity of D2, which could worsen gestational complications.

In the other hand, the TSHβ gene (NC_000001.11) located on chromosome 1 at position 38p12, codes for the beta unit of the thyroid stimulating hormone (TSH). It is admitted that genetic variants can show a different spectrum of actions.

This was a clinical, comparative, prospective and transversal study. Pregnant women aged 18-44 years old, were invited to identify it they had a DIO2 polymorphism or the TSHβX1 splice variant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attended at the "Mónica Pretelini Sáenz" Maternal-Perinatal Hospital (HMPMPS), Health Institute of the State of Mexico (ISEM), Toluca, Mexico.

Exclusion Criteria:

* Patients with chronic diseases other than hyper or hypothyroidism.
* Patients that required attention in the obstetric intensive care unit.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women attended at the "Mónica Pretelini Sáenz" Maternal-Perinatal Hospital are mainly of low socioeconomical status.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
TSHβX1 splice variant expression. | Baseline.
  Frequency of positive cases for the TSHβX1 splice variant identified by real-time polymerase change reaction.

SECONDARY OUTCOMES:
D2 Thr92Ala polymorphism. | Baseline.
  Allele frequency identification of the D2 Thr92Ala polymorphism by genotyping method.

CONTACTS AND LOCATIONS:
Overall Officials: Mendieta Zerón, Principal Investigator — Hospital Materno-Perinatal "Mónica Pretelini Sáenz".
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, Mexico

IPD SHARING:
Plan to Share IPD: No
The information will be available for academic journals if needed.

REFERENCES:
- [Background] Wouters HJ, van Loon HC, van der Klauw MM, Elderson MF, Slagter SN, Kobold AM, Kema IP, Links TP, van Vliet-Ostaptchouk JV, Wolffenbuttel BH. No Effect of the Thr92Ala Polymorphism of Deiodinase-2 on Thyroid Hormone Parameters, Health-Related Quality of Life, and Cognitive Functioning in a Large Population-Based Cohort Study. Thyroid. 2017 Feb;27(2):147-155. doi: 10.1089/thy.2016.0199. Epub 2016 Dec 15. PMID 27786042
- [Background] Leung AM. Thyroid function in pregnancy. J Trace Elem Med Biol. 2012 Jun;26(2-3):137-40. doi: 10.1016/j.jtemb.2012.03.004. Epub 2012 Jun 2. PMID 22658718
- See also: PREDICTED: Homo sapiens thyroid stimulating hormone beta (TSHB), transcript variant X1. — http://www.ncbi.nlm.nih.gov/nuccore/XM_011542065.2